CLINICAL TRIAL: NCT02422459
Title: Chronic Pain Self-Management Support With Pain Education and Exercise (COMMENCE): A Randomized Controlled Trial
Brief Title: Chronic Pain Self-management Support With Pain Education and Exercise
Acronym: COMMENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13-472
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COMMENCE (Experimental): ChrOnic pain self-ManageMent support with pain science EducatioN and exerCisE (COMMENCE)
  Interventions: Behavioral: COMMENCE
- Wait-list control (No Intervention): No treatment assigned

INTERVENTIONS:
Behavioral: COMMENCE — ChrOnic pain self-ManageMent support with pain science Education and exerCisE (COMMENCE) consists of two visits with a physiotherapist per week over six weeks. One of the two visits is in a group setting, where the emphasis is on pain neurophysiology education and provision of self-management strategies. The second visit each week is an individualized, one-to-one session in which the focus is on providing support for implementing self-management strategies and developing of an individualized, goal-oriented exercise program.
  Arms: COMMENCE

SUMMARY:
The purpose of this study is to determine whether the combination of self-management support, pain science education, and individualized, goal-oriented exercises helps people with chronic pain to increase their function.

DETAILED DESCRIPTION:
Primary objective: This study will test the hypothesis that participants with chronic pain experience greater change in function with ChrOnic pain self-ManageMent support with pain science EducatioN and exerCisE (COMMENCE) in comparison to a wait-list control.

Secondary objective #1: This study will test the hypotheses that people with chronic pain experience greater change in pain intensity, pain interference, self-efficacy, catastrophic thinking, fear of movement/re-injury, pain neurophysiology knowledge, how much participants are bothered by difficulty with functional activities, fatigue, depressive symptoms, health care utilization and work status with COMMENCE in comparison to a wait-list control.

Secondary objective #2: This study will identify demographic, psychological, or psychophysical variables that are predictive of treatment response.

Design: This study will be a randomized trial with parallel groups, a wait-list control and balanced randomization. A cross-over will take place after a 12-week follow-up assessment (ie. the group initially receiving treatment will receive no treatment and the group initially on the wait-list will receive treatment for 6 weeks). The between group comparison will be performed using only the data up to the 12-week follow-up due to anticipated carry-over effects with self-management support. Data collected after the cross-over will be used to help identify factors that predict response to the intervention.

Blinding: Due to the nature of the treatment and comparison, participants and the treating physiotherapist will not be blinded. The assessor who is completing the two objective measures will be blind to the treatment allocation. Data analysis will be performed by someone who is not blinded to the group allocation.

Setting: 110 participants with chronic pain will be recruited at Woodstock and Area Community Health Centre (WACHC) in Woodstock, Ontario, Canada. WACHC has an interdisciplinary team of health care providers that provide care to priority populations in Oxford County, Ontario, Canada. The priority populations include people with the following barriers to accessing health care: addictions concerns, mental health challenges, low incomes, lack of health insurance, and isolated seniors. The investigators expect this sample to represent a marginalized population of people with chronic often excluded from chronic pain treatment and research by barriers to accessing health care.

Sample Size: The sample size necessary for a randomized controlled trial with three repeated measures at 0, 7 and 18 weeks was calculated using online sample size software (GLIMMPSE 2.0). The calculation was performed using a significance level of 0.05, a power of 0.8, a minimum detectable mean difference between groups of 10 points on the Short Musculoskeletal Function Assessment Dysfunction Index (SMFA-DI) at both 7 weeks and 18 weeks, and a standard deviation of 23 points on the SMFA-DI based on clinical data at WACHC. The needed sample size calculated was 88 participants. To account for a potential 20% drop-out rate, 110 participants will be recruited

Allocation: The allocation sequence will be generated by a study investigator who is not involved in the enrolment of participants or assigning interventions. A computer-generated blocked random number schedule will be used to determine allocation sequence. The block size will be unknown to the other study investigators. The allocation sequence will be concealed through the use of sequentially numbered, opaque envelopes, opened after the initial assessment.

Co-intervention: Participants will be free to continue with other treatments. Other treatments will be recorded through self-report at each assessment time-point and analyzed for between group differences.

Withdrawing Participants from this Study: Participants may withdraw from the treatment at any time. Participants who choose to withdraw will be documented and data will be analyzed as a member of the group to which they were randomly assigned (intention-to-treat)

Potential prognostic indicators or predictors of response: Potential predictors of response for secondary objective #2 will include baseline measures for each of the outcome measures listed under outcomes as well as post-traumatic stress measured by the Post-traumatic Stress Disorder Checklist, sense of perceived injustice measured by the Injustice Experience Questionnaire, number of medications, comorbidities measured by disease count, and expectations for recovery. Expectations for recovery will be assessed with two questions: i) Do you think your pain will improve? ii) Do you think your functional abilities will improve?

Demographic information: The following information will be collected at the initial assessment and analyzed as potential covariates and predictors of response: age, sex, work status prior to symptom onset, length of time since symptom onset in months, diagnosis provided by a medical professional as reported by the patient, medication use, previous treatment received, and expectations for recovery.

Treatment fidelity: Treatment fidelity will be assessed through a combination of attendance (categorized as <25%, 25-49%, 50-74%, ≥75% of visits) and adherence to self-management strategies. This will be measured by clinician report when the clinician reviews the workbook at each individual treatment session.

Data monitoring and auditing: This trial will not include a data monitoring committee and will not be audited outside of the study investigators

Analysis: Statistical analysis will be conducted using Stata software, version 13 (StataCorp, College Station, Texas, USA). Baseline characteristics for treatment and wait-list groups will be compared using a Student's t-test for continuous data and Chi squared or Fisher's exact test for categorical variables. Analysis for the primary objective and secondary objective #1 will be performed using linear mixed-effects modelling with data from three repeated measures (baseline, 7 weeks, 18 weeks). A p value of less than 0.05 will be considered indicative of statistical significance. The primary analysis will use intention to treat principles, but a secondary analysis to investigate efficacy for those that complete 75% of visits will be performed as well (per protocol analysis). Predictors of response (change in SMFA-DI) will be determined using a series of multiple regression models.

ELIGIBILITY:
Inclusion Criteria:

* participants will all be adults who have been experiencing non-cancer related pain for at least 12 weeks

Exclusion Criteria:

* cancer related pain
* medical "red flags" suggestive of a non-neuromusculoskeletal etiology of symptoms
* casted fracture within the last 12 weeks
* related surgery within the last 26 weeks
* evidence of upper motor neuron lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Short-Musculoskeletal Function Assessment - Dysfunction Index | change in function from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  Measures function

SECONDARY OUTCOMES:
Short-Musculoskeletal Function Assessment - Bother Index | change in bother index from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures how much participants are bothered by difficulty completing functional activities
Numeric Pain Rating Scale | change in pain intensity from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures pain intensity
PROMIS Pain Interference Item-Bank - 8 Items | change in pain interference from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures pain interference
Numeric Fatigue Rating Scale | change in fatigue from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures fatigue
Patient Health Questionnaire - 9 | change in depressive symptoms from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures depressive symptoms
Pain Catastrophizing Scale | change in catastrophizing from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures catastrophic thinking related to pain
Tampa Scale of Kinesiophobia - 11-item | change in fear of movement/re-injury from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures fear of movement/re-injury
Pain Self-Efficacy Questionnaire | change in self-efficacy from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures self-efficacy
Neurophysiology of Pain Questionnaire - Revised | change in knowledge from baseline at 18 weeks (12 week follow-up) with repeated measures at 0, 7 and 18 weeks
  measures participants knowledge of pain neurophysiology
Number of health care visits over 12 weeks | change in number of health care visits from 12-weeks immediately prior to treatment to number of visits during 12-week follow-up period
  Measures health care utilization
Work status | Change in work status from baseline at 18 weeks
  measure of vocational participation
Number of visits attended | Number of visits during 6 week treatment period
  measure of treatment fidelity
Adverse events or harms reported | Number of adverse events reported during 6 week treatment period
  Measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD(c), Principal Investigator — McMaster University; Joy C MacDermid, PhD, Principal Investigator — McMaster University
Locations (1):
- Woodstock and Area Community Health Centre, Woodstock, Ontario, Canada

REFERENCES:
- [Derived] Miller J, MacDermid JC, Walton DM, Richardson J. Chronic Pain Self-Management Support With Pain Science Education and Exercise (COMMENCE) for People With Chronic Pain and Multiple Comorbidities: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 May;101(5):750-761. doi: 10.1016/j.apmr.2019.12.016. Epub 2020 Jan 29. PMID 32004517
- [Derived] Miller J, MacDermid JC, Walton DM, Richardson J. Chronic pain self-management support with pain science education and exercise (COMMENCE): study protocol for a randomized controlled trial. Trials. 2015 Oct 14;16:462. doi: 10.1186/s13063-015-0994-5. PMID 26466908